CLINICAL TRIAL: NCT01291758
Title: Exercise in Gulf War Illness (GWI)
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, James Baraniuk, MD, Professor of Medicine, Georgetown University
Other Study IDs: 2009-229; USAMRMC PR# W81XWH-09-1-0526 (Other Grant/Funding Number: Department of Defense); HRPO Log No. A-15547 (Other: Human Research Protection Office)
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Gulf War Illness; Persian Gulf Syndrome
Keywords: Persian Gulf War; Gulf War Syndrome; GWI; Gulf War Illness; Exercise; Chronic Fatigue; Fibromyalgia; Veterans; Irritable Bowel Syndrome; Migraine headaches; Neuropathy
MeSH Terms: conditions — Persian Gulf Syndrome; Motor Activity; Fibromyalgia; Irritable Bowel Syndrome; Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum, urine, cerebrospinal fluid (CSF), and buccal swab samples retained for testing as described in protocol.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- GWI: Veterans of the 1990-1991 Persian Gulf War who have autonomic, neurological and other symptoms
  Interventions: Diagnostic Test: Submaximal bicycle exercise stress tests performed 24 hr apart
- HC: Healthy veterans of the 1990-1991 Persian Gulf War
  Interventions: Diagnostic Test: Submaximal bicycle exercise stress tests performed 24 hr apart

INTERVENTIONS:
Diagnostic Test: Submaximal bicycle exercise stress tests performed 24 hr apart — Submaximal bicycle exercise stress tests were performed for 25 min at 70% predicted heart rate, then ramped up to 85% predicted heart rate. Subjects could stop when they felt they had reached their maximum effort if before reaching 85% predicted heart rate.

SUMMARY:
The purpose of this study is to determine if submaximal exercise by bicycle stress tests with pulmonary measurement of VO2MAX plus maximal isometric hand grips on 2 consecutive days causes a higher level of "exertional exhaustion" in GWI compared to healthy veterans (HVets).

DETAILED DESCRIPTION:
Subjects sat on upright bicycles for preexercise symptoms, respiratory gases, EKG, and vital sign measurements.

Submaximal exercise began at low resistance with increases every 30 to 60 seconds until 70% predicted heart rate was reached by 5 minutes. Subjects maintained their pace until 25 minutes, then resistance was increased incrementally to increase to 85% predicted heart rate (approximately sufficient to reach anaerobic threshold).

Symptoms, respiratory gases, EKG, and vital signs were measured every 5 minutes, at peak of exercise, and 5 minute intervals after exercise.

The identical exercise protocol was used approximately 24 hr later. Secondary outcomes were assessed by comparisons from before exercise to after the second bicycle exercise stress test.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of military enlistment between August 1, 1990 and July 31, 1991, and deployment for 30 consecutive days to:

  * Persian Gulf waters and adjacent land areas
  * Other global locations
  * U.S. only
* Status prior to 1990 and 1991:

  * Active duty
  * National Guard
  * Reserves

Exclusion Criteria:

* Current active duty military personnel
* Any one who was not active duty military personnel between August 1, 1990 and July 31, 1991
* HIV/AIDS; pregnancy or lactation; potential hepatitis; drug addiction; chronic inflammatory, infectious, or autoimmune medical illnesses not associated with GWI; incarceration; dementia, other cognitive limitation; or reliance on a care-giver in order to respond to the questionnaires and other study tests.

Amputations of one or both hands and forearms will be permitted but hand grip tests will not be tested

Ages: 38 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All veterans who served in the Armed Forces between August 1990 and July 1991
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
To assess the alterations due to exercise in Gulf War Veterans | 02/2009-09/2012
  Difference in duration of exercise between first and second submaximal bicycle exercise stress test

CONTACTS AND LOCATIONS:
Overall Officials: James N Baraniuk, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Contact James N. Baraniuk MD at baraniuj@geogetown.edu Each request will be reviewed by Dr. Baraniuk and may require approval from the Georgetown University IRB Committee before data can be shared.
  Efforts are underway to deidentify data for public access.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data are available for collaborative research as in Plan Description.
Access Criteria: Access depends on the request and need for IRB approval

REFERENCES:
- [Background] Gray GC, Reed RJ, Kaiser KS, Smith TC, Gastanaga VM. Self-reported symptoms and medical conditions among 11,868 Gulf War-era veterans: the Seabee Health Study. Am J Epidemiol. 2002 Jun 1;155(11):1033-44. doi: 10.1093/aje/155.11.1033. PMID 12034582
- [Background] Baraniuk JN, Casado B, Maibach H, Clauw DJ, Pannell LK, Hess S S. A Chronic Fatigue Syndrome - related proteome in human cerebrospinal fluid. BMC Neurol. 2005 Dec 1;5:22. doi: 10.1186/1471-2377-5-22. PMID 16321154
- [Background] Janssen B, Hohenadel D, Brinkkoetter P, Peters V, Rind N, Fischer C, Rychlik I, Cerna M, Romzova M, de Heer E, Baelde H, Bakker SJ, Zirie M, Rondeau E, Mathieson P, Saleem MA, Meyer J, Koppel H, Sauerhoefer S, Bartram CR, Nawroth P, Hammes HP, Yard BA, Zschocke J, van der Woude FJ. Carnosine as a protective factor in diabetic nephropathy: association with a leucine repeat of the carnosinase gene CNDP1. Diabetes. 2005 Aug;54(8):2320-7. doi: 10.2337/diabetes.54.8.2320. PMID 16046297
- [Background] Casado B, Zanone C, Annovazzi L, Iadarola P, Whalen G, Baraniuk JN. Urinary electrophoretic profiles from chronic fatigue syndrome and chronic fatigue syndrome/fibromyalgia patients: a pilot study for achieving their normalization. J Chromatogr B Analyt Technol Biomed Life Sci. 2005 Jan 5;814(1):43-51. doi: 10.1016/j.jchromb.2004.09.056. PMID 15607706
- [Background] Fukuda K, Nisenbaum R, Stewart G, Thompson WW, Robin L, Washko RM, Noah DL, Barrett DH, Randall B, Herwaldt BL, Mawle AC, Reeves WC. Chronic multisymptom illness affecting Air Force veterans of the Gulf War. JAMA. 1998 Sep 16;280(11):981-8. doi: 10.1001/jama.280.11.981. PMID 9749480
- [Result] Rayhan RU, Zheng Y, Uddin E, Timbol C, Adewuyi O, Baraniuk JN. Administer and collect medical questionnaires with Google documents: a simple, safe, and free system. Appl Med Inform. 2013;33(3):12-21. PMID 24415903
- [Result] Rayhan RU, Ravindran MK, Baraniuk JN. Migraine in gulf war illness and chronic fatigue syndrome: prevalence, potential mechanisms, and evaluation. Front Physiol. 2013 Jul 24;4:181. doi: 10.3389/fphys.2013.00181. eCollection 2013. PMID 23898301
- [Result] Rayhan RU, Stevens BW, Raksit MP, Ripple JA, Timbol CR, Adewuyi O, VanMeter JW, Baraniuk JN. Exercise challenge in Gulf War Illness reveals two subgroups with altered brain structure and function. PLoS One. 2013 Jun 14;8(6):e63903. doi: 10.1371/journal.pone.0063903. Print 2013. PMID 23798990
- [Result] Rayhan RU, Stevens BW, Timbol CR, Adewuyi O, Walitt B, VanMeter JW, Baraniuk JN. Increased brain white matter axial diffusivity associated with fatigue, pain and hyperalgesia in Gulf War illness. PLoS One. 2013;8(3):e58493. doi: 10.1371/journal.pone.0058493. Epub 2013 Mar 20. PMID 23526988
- [Derived] Narayan V, Shivapurkar N, Baraniuk JN. Informatics Inference of Exercise-Induced Modulation of Brain Pathways Based on Cerebrospinal Fluid Micro-RNAs in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome. Netw Syst Med. 2020 Nov 18;3(1):142-158. doi: 10.1089/nsm.2019.0009. eCollection 2020. PMID 33274349
- See also: Laboratory Website — http://www9.georgetown.edu/faculty/baraniuj/Site/Welcome.html